CLINICAL TRIAL: NCT06058546
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase II Clinical Trial of Efficacy and Safety of Jiuweihuaban Pill in the Treatment of Moderate to Severe Plaque Psoriasis(Syndrome of Blood-heat ).
Brief Title: Efficacy and Safety of Jiuweihuaban Pill for Treating Plaque Psoriasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-JWHBW-II
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Jiuweihuaban Pill placebo, 1 bag each time, p.o. , tid
  Interventions: Drug: Jiuweihuaban Pill placebo
- Low dose group (Experimental): Jiuweihuaban Pill , 1 bag each time, p.o. , tid
  Interventions: Drug: low dose Jiuweihuaban Pill
- High dose group (Experimental): Jiuweihuaban Pill , 1 bag each time, p.o. , tid
  Interventions: Drug: high dose Jiuweihuaban Pill

INTERVENTIONS:
Drug: Jiuweihuaban Pill placebo — Jiuweihuaban pill placebo 1 bag(12 g placebo per bag),p.o.,tid,for 12weeks.
  Other Names: Placebo group
  Arms: Placebo group
Drug: low dose Jiuweihuaban Pill — Low dose Jiuweihuaban pill 1 bag(3 g placebo per bag and 9 g Jiuweihuaban pill ),p.o.,tid,for 12weeks.
  Other Names: Low dose group
  Arms: Low dose group
Drug: high dose Jiuweihuaban Pill — High dose Jiuweihuaban pill 1 bag(12 g Jiuweihuaban pill ),p.o.,tid,for 12weeks.
  Other Names: High dose group
  Arms: High dose group

SUMMARY:
This study will evaluate the efficacy and safety of Jiuweihuaban Pill in the treatment of moderate to severe plaque psoriasis(syndrome of blood-heat ).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65, male or female.
2. The diagnosis of plaque psoriasis vulgaris was in accordance with the western diagnostic criteria
3. Conformed to the TCM syndrome differentiation standard of plaque psoriasis with Blood-heat syndrome.
4. At screening period: 3 ≤PASI≤ 20, 3%≤BSA≤ 10% and sPGA≥2.
5. Willing to participate voluntarily and sign a written informed consent.

Exclusion Criteria:

1. Psoriasis caused by drug-induced factors; combined with non-plaque Psoriasis at screening (such as guttate,arthropathica, pustular, erythrodermic and other types of Psoriasis); The skin lesions are exclusively observed in subjects with specific areas such as the face, scalp, nails, skin folds, glans penis, mucous membranes, palms, and soles.
2. Systemic therapy with non-biological drugs within 4 weeks prior to randomization, including but not limited to systemic corticosteroids, retinoids, methotrexate, and cyclosporine.
3. Systemic therapy with biological drugs within 12 weeks or 5 half-lives (whichever is longer) prior to randomization, including but not limited to interleukin antibodies (such as ustekinumab, secukinumab) and tumor necrosis factor-alpha antagonists (such as etanercept, infliximab, adalimumab) in the study.
4. Topical anti-psoriatic treatment received within 2 weeks prior to randomization, including retinoids, vitamin D3 derivatives, corticosteroids, and others
5. Physical therapy received within the 4 weeks prior to randomization, including phototherapy (such as UVB, PUVA), combination phototherapy, and balneotherapy.
6. Systemic anti-infective treatment received within the 4 weeks prior to randomization; presence of recurrent, chronic, or active infection at baseline as determined by the investigator and judged to increase the subject's risk.
7. With a serious, progressive, or uncontrolled disease, including but not limited to a disease of the immune (such as rheumatoid arthritis, systemic lupus erythematosus, and inflammatory bowel disease), endocrine, hematological, urinary, hepatobiliary, and respiratory, nervous, psychiatric, cardiovascular, gastrointestinal, or infectious system, a malignancy.
8. Patients with serum creatinine above the upper limit of normal at screening, with elevated Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) levels ≥ 1.5 times the upper limit of normal.
9. Participation in other clinical trials and received investigational drugs within 1 month prior to screening.
10. Patients with hypersensitivity to the investigational drug components.
11. Patients had a history of smoking, alcohol, drug abuse.
12. Patients (including partners) have plans to become pregnant from 2 weeks before the first dose to 1 month after the last dose and Subjects do not take effective contraceptive measures during this period or during pregnancy or breastfeeding
13. Any other situation that the investigator did not consider suitable for participation in the study, such as other skin problems that hinder the assessment of Psoriasis, potential compliance problems, inability to complete all examinations and evaluations in accordance with the protocol requirements, may pose an uncontrollable risk for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
PASI 75 | Baseline to days 84.
  Proportion of subjects achieving an improvement of ≥75% in Psoriasis Area and Severity Index (PASI75) from baseline at days84.

SECONDARY OUTCOMES:
PASI75 | Baseline to days 28、56.
  Proportion of subjects achieving an improvement of ≥75% in Psoriasis Area and Severity Index (PASI75) from baseline at days 28、56.
PASI50、90 | Baseline to days 28、56、84.
  Proportion of subjects achieving an improvement of ≥50% and ≥90% in Psoriasis Area and Severity Index (PASI50, PASI90) from baseline at days 28、56、84.
Change value and percentage change in PASI score | Baseline to days 84.
  Change value and percentage change in PASI score from baseline at days 84.The PASI scores can range from 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0, corresponding to maximal signs of psoriasis.
Proportion of subjects achieving sPGA=0 or 1 | Baseline to days 28、56、84.
  Proportion of subjects achieving clear (score of 0) or almost clear (score of 1) in static Physician Global Assessment (sPGA=0 or 1) at Weeks 4, 8, and 12.
Proportion of subjects achieving an improvement of ≥2 points in sPGA | Baseline to days 28、56、84.
  Proportion of subjects achieving an improvement of ≥2 points in static Physician Global Assessment from baseline at days 28、56、84.
Change value and percentage change in BSA affected by psoriasis | Baseline to days 28、56、84.
  Change value and percentage change in Body Surface Area (BSA) affected by psoriasis from baseline at days 28、56、84.
Change value and percentage change in NRS for skin itching | Baseline to days 28、56、84.
  Change value and percentage change in Numeric Rating Scale (NRS) for skin itching from baseline at days 28、56、84. The NRS scores can range from 0,corresponding to no itching symptom，up to a maximum of 10,corresponing to the most severe itching .
Change value and percentage change in DLQI score | Baseline to days 28、56、84.
  Change value and percentage change in Dermatology Life Quality Index (DLQI) score from baseline at days 28、56、84. The DLQI scores can range from 0 to 30.The higher the score, the worse the quality of life.
Proportion of subjects achieving DLQI=0-1 | Baseline to days 28、56、84.
  Proportion of subjects achieving a DLQI score of 0-1 (DLQI=0-1) at days 28、56、84.The DLQI scores can range from 0 to 30.The higher the score, the worse the quality of life.
Change value and percentage change in Traditional Chinese Medicine Syndrome score | Baseline to days 28、56、84.
  Change value and percentage change in Traditional Chinese Medicine Syndrome score from baseline at days 28、56、84.The Traditional Chinese Medicine Syndrome scores can range from 0 to 27.The higher the score, the more severe psoriasis.
Disappearance rate of individual symptoms in Traditional Chinese Medicine Syndrome | Baseline to days 28、56、84.
  Disappearance rate of individual symptoms in Traditional Chinese Medicine Syndrome at days 28、56、84.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing traditional Chinese medicine hospital affiliated to Capital Medical University, Beijing
  - Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun
  - The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha
  - Chengdu Second People's Hospital, Chengdu
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan
  - Yunnan Provincial Hospital of Traditional Chinese Medicine, Kunming
  - Nanyang First People's Hospital, Nanyang
  - The First Affiliated Hospital of China Medical University, Shenyang
  - Affiliated Hospital of Tianjin Institute of Traditional Chinese Medicine, Tianjin
  - First affiliated hospital of Wenzhou medical university, Wenzhou
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen
  - Xingtai people's hospital, Xingtai